CLINICAL TRIAL: NCT00590928
Title: Effect of Intravenous Esomeprazole Versus Ranitidine on Gastric pH in Critically Ill Patients - a Prospective, Randomized, Double-Blind Study.
Brief Title: Gastric pH in Critically Ill Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Christian Madl, MD, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13H1-CM1; ESORAN trail
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Last update posted 2008-01-11 (Estimated); Status verified 2007-12

CONDITIONS: Critically Ill Patients; Indication for Stress Ulcer Prophylaxis
MeSH Terms: interventions — Esomeprazole; Ranitidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): patients with indication for stress ulcer prophylaxis and gastric pH < 4
  Interventions: Drug: esomeprazole
- 2 (Active Comparator): patients with indication for stress ulcer prophylaxis and gastric pH < 4
  Interventions: Drug: ranitidine

INTERVENTIONS:
Drug: esomeprazole — 40mg once daily
  Arms: 1
Drug: ranitidine — 50mg every h hours
  Arms: 2

SUMMARY:
H2-receptor antagonists are the gold standard for stress ulcer prophylaxis in critically ill patients. Various studies demonstrated superiority of proton pump inhibitors over H2-receptor antagonists in increasing gastric pH and in healing gastric acid-dependent diseases. It is unknown, whether proton pump inhibitors are more effective in increasing gastric pH than H2-receptor antagonists in critically ill patients requiring stress ulcer prophylaxis.

DETAILED DESCRIPTION:
Gastric pH is measured continuously for 72 hours with a pipolar microelectrode placed between 7 and 15cm below the lower esophageal sphincter.

ELIGIBILITY:
Inclusion Criteria:

* critically ill patients
* indication for stress ulcer prophylaxis
* gastric pH < 4

Exclusion Criteria:

* gastrointestinal bleeding
* gastric pH > 4

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2004-07; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
the percentage of time with gastric pH > 4 | 72 hours

SECONDARY OUTCOMES:
median gastric pH | 72 hours
incidence of gastrointestinal bleeding | 72 hours
incidence of ventilator associated pneumonia | ICU stay
the percentage of time with an gastric pH > 5 | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Christian Madl, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Department of Medicine III, ICU, Vienna, Austria